CLINICAL TRIAL: NCT05447975
Title: A Prospective Cohort Study of Exercise Rehabilitation in the Treatment of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shengdi Chen, Professor, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RuijinH-202205
Record Dates: First submitted 2022-05-27; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi group (Experimental)
  Interventions: Other: Tai Chi training
- Control (No Intervention)

INTERVENTIONS:
Other: Tai Chi training — As for Tai Chi training, standardized Tai Chi was taught by professional Tai Chi coaches from Sino Taiji of Fuxing International in classes: Qishi ("Starting Posture"), Shangsanbu ("Twist Step"), Yema Fenzong("Part the Wild Horse's Mane on Both Side"), Jingang Daozhui ("Buddha's warrior attendant pounds mortar"), Shoushi ("Closing Posture"). Patients participated in this class were trained, twice a week, 60 min per time. PD patients whose attendance rate less than 75% were excluded.
  Arms: Tai Chi group

SUMMARY:
The investigators proposed to conduct a cohort study to observe whether Tai Chi intervention could delay the disease progression of Parkinson's disease (PD).

PD patients were enrolled into 5 Tai Chi classes which began at different timepoints from Jan. 2016 to Jan. 2019. Each participant was assessed before participants joined the Tai Chi class. After the recruitment, participants accepted continuous Tai Chi training in the classes till the last follow-up. The investigators performed three times of follow-up in Nov. - Dec. 2019, Oct. - Nov. 2020 and Jun. - July 2021. Using propensity score matching, the investigators matched PD patients who did not receive Tai Chi training as control group in gender, disease duration, age, and Hoehn - Yahr staging. The aim is to observe the effect of Tai Chi on delaying the disease progression of PD.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Parkinson's disease according to 2015 MDS diagnostic criteria and United Kingdom Brain Bank diagnostic criteria in 1992;
2. Hoehn - Yahr staging: 1 - 2.5;
3. The medication was stable at least 3 months before recruiting and not changed during follow-up unless increasing antiparkinsonian drugs or the need of deep brain stimulation (DBS) is required according to the disease severity;

Exclusion Criteria:

1. Secondary causes, such as inflammatory, drug-induced, vascular and toxin-induced parkinsonism.
2. Parkinsonism with other neurodegenerative diseases, such as progressive supranuclear palsy, multiple system atrophy, cortical basal ganglia degeneration, Wilson's disease.
3. Other neurological diseases, such as stroke.
4. Patients who were receiving any other clinical trials or regular exercise protocols.
5. Patients who had fall incidents in the 6 months before recruiting due to safety considerations.
6. Patients whose Mini-Mental State Examination (MMSE) scores were less than 24.
7. Patients who had medical history that did not fit to exercise, such as orthopedics diseases or cardiopulmonary dysfunction.
8. Patients who received education less than 6 years.
9. Patients who could not walk and live independently.
10. Patients who received brain surgery (e.g. deep brain stimulation);
11. Patients whose exercise length longer than 50 minutes per week.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
the annual change of UPDRS total score measured in "ON" state at three follow-ups | 1 year
  the annual change of Unified Parkinson's Disease Rating Scale (UPDRS) total score measured in "ON" state at three follow-ups. The range of UPDRS is between 0 and 207. The higher score means a worse outcome.

REFERENCES:
- [Derived] Li G, Huang P, Cui S, He Y, Tan Y, Chen S. Effect of long-term Tai Chi training on Parkinson's disease: a 3.5-year follow-up cohort study. J Neurol Neurosurg Psychiatry. 2024 Feb 14;95(3):222-228. doi: 10.1136/jnnp-2022-330967. PMID 37875337

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT05447975/Prot_SAP_000.pdf